CLINICAL TRIAL: NCT01583192
Title: Prospective Study of Chloridehexidine/Alcohol Versus Jodine/Povidine in Forefoot Surgery
Brief Title: Chloridehexidine Versus Povidine Jodine Both Soluted in Alcohol in Forefoot Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Mario Speth, MD, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: mbshadid
Record Dates: First submitted 2012-03-23; First posted 2012-04-23 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Hallux Valgus; Arthritis of the First Metatarsophalangeal Joint
Keywords: infection; skin preparation; fore-foot surgery; chloride-hexidine; povidine-jodine; alcohol
MeSH Terms: conditions — Hallux Valgus; Infections | interventions — Skin Lightening Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- chloride-hexidine soluted in alcohol (Active Comparator): patients will have skin preparation with chloride-hexidine soluted in alcohol prior to their forefoot surgery.
  Skin swabs will be taken prior to skin preparation, after skin preparation and after skin closure at the end of the operation
  Interventions: Procedure: skin preparation
- povidine-jodine soluted in alcohol (Active Comparator): skin perparation will be done with povidine-jodine soluted in alcohol prior to forefoot surgery.
  Interventions: Procedure: skin preparation

INTERVENTIONS:
Procedure: skin preparation — skin preparation while be done either with chloride-hexidine 0,5% soluted in alcohol 70% or povidine-jodine 1% soluted in alcohol 70%

SUMMARY:
The study will prospectively compare the efficacy and safety of chloride hexidine soluted in alcohol with povidine-jodine soluted in alcohol in forefoot surgery.

DETAILED DESCRIPTION:
It will be a comparative study in which we will swab cultures before skin preparation directly after skin preparation and at the and of the operation (hallux valgus correction and arthrodesis of the first metatarsophalangeal joint.

There will be a quantitative and quality analysis of the swabs. We will also measure allergic reactions. During the post-operative period of 6 weeks we will measure the wound infections stated by Prezies.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years
* written informed consent
* indication for hallux valgus correction or arthrodesis of the first metatarsophalageal joint

Exclusion Criteria:

* allergic for jodine-povidine and/or chloride-hexidine
* active infection
* skin defect
* blood clotting or coagulation disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
number of positive swab cultures | From start surgery week until 48 hours post-operatively
  During surgery swabs will be taken before skin desinfection, after skin desinfection and at the end of the surgery.
  We will count the number of positive swab cultures taken from the webspace of their first and second toe and at the place of incision 48 hours post-operatively.
wound infection | until 6 weeks postoperatively
  we will count the number of wound infections, stated by Prezies, for a period of 6 weeks postoperatively

SECONDARY OUTCOMES:
Allergic events | Until 6 weeks postoperatively
  we will look at the number of allergic events occuring.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Speth, MD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St Antonius Hospital, Nieuwegein, Utrecht, Netherlands

REFERENCES:
- See also: woundinfection criteria — http://www.prezies.nl/zkh/definities/Definities_POWI_2012.pdf